CLINICAL TRIAL: NCT05728294
Title: Femoral or Sciatic Nerve Block to Provide Analgesia After Proximal Tibial Osteotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Program Director, regional anaesthesia, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-01774
Record Dates: First submitted 2023-01-19; First posted 2023-02-15 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Two groups: femoral nerve block or sciatic nerve block with ropivacaine
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Femoral nerve block (Active Comparator): Femoral nerve block performed under ultrasound guidance with ropivacaine 0.5%, 20mL
  Interventions: Procedure: Femoral nerve block with ropivacaine 0.5%, 20 ml
- Sciatic nerve block (Experimental): Sciatic nerve block performed under ultrasound guidance with ropivacaine 0.5%, 20mL
  Interventions: Procedure: Sciatic nerve block with ropivacaine 0.5%, 20 ml

INTERVENTIONS:
Procedure: Femoral nerve block with ropivacaine 0.5%, 20 ml — Femoral nerve block under ultrasound guidance with ropivacaine 0.5%, 20 ml
  Arms: Femoral nerve block
Procedure: Sciatic nerve block with ropivacaine 0.5%, 20 ml — Sciatic nerve block under ultrasound guidance with ropivacaine 0.5%, 20 ml
  Arms: Sciatic nerve block

SUMMARY:
Proximal tibial osteotomy is associated with moderate to severe postoperative pain. The proximal part of the tibia is innervated by branches from the femoral nerve anteriorly and the sciatic nerve posteriorly. Little is known on the type of peripheral nerve block to perform so that optimal postoperative analgesia is provided with minimum impact on the motor function. This randomised controlled double-blinded trial tested the hypothesis that a femoral nerve block provides superior analgesia than a sciatic nerve block after proximal tibial osteotomy.

ELIGIBILITY:
Inclusion Criteria:

* proximal tibial osteotomy

Exclusion Criteria:

* femoral or sciatic nerve deficit,
* pre-existing peripheral neuropathy,
* chronic pain diagnosis,
* pregnancy,
* identified contraindications to peripheral nerve block (e.g., local anesthetic allergy, coagulopathy, or infection at the block site).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Intravenous morphine consumption | 24 hours after surgery
  Intravenous morphine consumption (mg)

SECONDARY OUTCOMES:
Intravenous morphine consumption | 2 hours after surgery
  Intravenous morphine consumption (mg)
Intravenous morphine consumption | 48 hours after surgery
  Intravenous morphine consumption (mg)
rest pain score | 2 hours after surgery
  pain score at rest (visual analogue scale, 0-10)
rest pain score | 24 hours after surgery
  pain score at rest (visual analogue scale, 0-10)
rest pain score | 48 hours after surgery
  pain score at rest (visual analogue scale, 0-10)
dynamic pain score | 2 hours after surgery
  pain score on movement (visual analogue scale, 0-10)
dynamic pain score | 24 hours after surgery
  pain score on movement (visual analogue scale, 0-10)
dynamic pain score | 48 hours after surgery
  pain score on movement (visual analogue scale, 0-10)
Rate of postoperative nausea and vomiting | 2 hours after surgery
  number of events/total number of patients
Rate of postoperative nausea and vomiting | 24 hours after surgery
  number of events/total number of patients
Rate of postoperative nausea and vomiting | 48 hours after surgery
  number of events/total number of patients

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Lausanne, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Kull C, Martin R, Rossel JB, Nguyen A, Albrecht E. Femoral vs sciatic nerve block to provide analgesia after medial open wedge high tibial osteotomy in the setting of multimodal analgesia: A randomized, controlled, single-blinded trial. J Clin Anesth. 2024 May;93:111355. doi: 10.1016/j.jclinane.2023.111355. Epub 2023 Dec 21. PMID 38134484